CLINICAL TRIAL: NCT01417819
Title: Effect of a Mobile Phone Short Message Service (SMS) on Childhood Cataract Follow-up Adherence in China
Brief Title: Effect of Mobile Communication on Childhood Cataract Follow-up Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CCPMOH2010-China1
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SMS reminder (Other): SMS reminders four days and one day before their appointments
  Interventions: Other: Mobile short message service

INTERVENTIONS:
Other: Mobile short message service — Mobile short message service reminder for appointments of parents of cataract children
  Other Names: Fetion, China Mobile

SUMMARY:
Rigorous and regular follow-up is essential to successful management of childhood cataract, but it is often ignored by parents and especially difficult to be delivered in China, such an average-medical-resource-limited country.

Health programmes that use mobile communication technologies are emerging with the aim of strengthening health systems.

The investigators aimed to assess whether mobile phone short message service (SMS) for parents of cataract children involved in the Childhood Cataract Program of Ministry of Health of China (CCPMOH) improved follow-up adherence and detection rate of the timing of surgery, postoperative complications and necessary replacement of glasses.

DETAILED DESCRIPTION:
Congenital and developmental cataract is a priority of Vision 2020: the Right to Sight, the global initiative to reduce the world's burden of avoidable blindness, because it is an important treatable cause of visual handicap in childhood throughout the world. Successful management of childhood cataract is dependent on early diagnosis and referral for surgery when indicated. Accurate optical rehabilitation and postoperative supervision are also essential. The timing of surgery of childhood cataract depends on the etiology and on the degree of visual interference. Severe bilateral cataracts with significant obstruction of the visual axis must be treated and surgery is recommended as soon as possible after discovery. Ideally cataracts should be removed before 3 months of age. In unilateral congenital cataract cases the prognosis for useful vision following surgery depends on prompt restoration of a clear visual axis, correction of aphakia, and aggressive treatment of amblyopia. In China, severe visual impairment is common in pediatric patients with cataract, and delayed presentation to hospital and late surgical treatment are found to be the major reasons. Therefore, in order to control childhood blindness and severe visual impairment in China, it is essential to ensure that pediatric patients with cataract could have good timing of surgery, postoperative rigorous supervision, accurate optical rehabilitation and aggressive treatment of amblyopia.

The importance of follow-up has been widely accepted and applied for research by many clinical disciplines. It is no doubt that rigorous and regular follow-up is essential to successful management of childhood cataract, for the cataract degree and visual development are individually different and changing, and the long-term visual acuity might be influenced by many factors. In other word, individual strategy according to the results of follow-up is the best choice for management of childhood cataract. The key to make the most appropriate individual strategy for each cataract child is strict follow-up on the basis of good communication. However, communicating with children and their families is complex, routinely involves the physician-parent-child triad and other family members, and is influenced by the developmental and cognitive stage of the child, interaction dynamics within the family, and differing parent and child needs. In addition to communication difficulties, financial difficulty and transportation difficulties were also the common causes for pediatric patients' parents to refusal or abandonment of treatment plan in China.

As a developing country, China's health-care level is currently unsatisfactory and the health-care reform still needs a long way to go. However, with the rapid economic development, Chinese cell phone users exceed 900 million people and this amount is to make China as a country with the largest number of mobile phone users in the world, mainly because of huge population and economic development, without factors related to healthcare. Actually, mobile phone communication has been suggested as a method to improve delivery of health services around the world, and most of the researches of health care via mobile phone are focused on HIV/AIDS, tuberculosis, and malaria. As an average-medical-resource-limited country but the largest mobile phone market, China should more use the potential of mobile technology in health systems compared to other countries. It is one of the goals of health-care reform that a wide range of medical services could be improved by providing patient-focused support and management through the health-care system. If mobile phone use does improve health outcomes in resource-limited settings, especially for chronic, congenital and developmental diseases needing good communication and collaboration, such as childhood cataract, this mobile health technology could thus be included in health-system strategies and help improve health development goals.

In this trial, we aimed to assess whether mobile phone communication between pediatric ophthalmologists and parents of cataract children involved in the Childhood Cataract Program of Ministry of Health of China improved follow-up adherence and detection rate of the timing of surgery, postoperative complications and necessary replacement of glasses.

ELIGIBILITY:
Inclusion Criteria:

* If the children were identified with congenital or development cataract before or after surgery, without other ocular abnormality
* Parents were able to access a mobile phone on a near-daily basis and communicate via short message service (SMS).
* Have signed a consent form
* Can be followed

Exclusion Criteria:

* Children not identified with congenital or development cataract
* Parents without ownership of mobile phone
* Have not signed consent form
* Be not able to be followed

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 258 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
follow-up adherence | up to 24 weeks
  Follow-up adherence included the rates of attendance, non-attendance, and rates of several categories of attrition (withdrawal from the study, transfer to non-study clinics, and loss to follow-up without identifiable cause).

SECONDARY OUTCOMES:
necessary management rates | up to 24 weeks
  Including:Surgery rates,laser treatment rates,replacement rates of glasses and incidence of secondary glaucoma

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Cheng, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen U, Guangzhou, Guangdong, China

REFERENCES:
- [Background] You C, Wu X, Zhang Y, Dai Y, Huang Y, Xie L. Visual impairment and delay in presentation for surgery in chinese pediatric patients with cataract. Ophthalmology. 2011 Jan;118(1):17-23. doi: 10.1016/j.ophtha.2010.04.014. Epub 2010 Aug 14. PMID 20709402
- [Background] Chak M, Wade A, Rahi JS; British Congenital Cataract Interest Group. Long-term visual acuity and its predictors after surgery for congenital cataract: findings of the British congenital cataract study. Invest Ophthalmol Vis Sci. 2006 Oct;47(10):4262-9. doi: 10.1167/iovs.05-1160. PMID 17003414
- [Background] Rider EA, Volkan K, Hafler JP. Pediatric residents' perceptions of communication competencies: Implications for teaching. Med Teach. 2008;30(7):e208-17. doi: 10.1080/01421590802208842. PMID 18777421
- [Background] Padma TV. Developing solutions. Nature. 2010 Jul 15;466(7304):S16-7. doi: 10.1038/nature09242. No abstract available. PMID 20631698
- [Background] Krishna S, Boren SA, Balas EA. Healthcare via cell phones: a systematic review. Telemed J E Health. 2009 Apr;15(3):231-40. doi: 10.1089/tmj.2008.0099. PMID 19382860
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Derived] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- See also: Home page of ZHONGSHANG OPHTHALMIC CENTER — http://www.gzzoc.com/
- See also: Home of Cataract Children — http://www.cnccclub.com/